CLINICAL TRIAL: NCT06730828
Title: Use of Amiodarone-Infused CardiaMend (CardiaMend-Amiodarone) Patches for the Prevention of New-Onset Postoperative Atrial Fibrillation (POAF) in Subjects Undergoing Cardiac Surgery
Brief Title: Amiodarone-Infused CardiaMend Patches for the Prevention of New-Onset POAF in Cardiac Surgery Subjects
Acronym: AMIOMEND
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Helios Cardio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP001
Record Dates: First submitted 2024-12-03; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation, Postoperative
Keywords: post Operative Atrial Fibrillation; Arrhythmias; Cardiac Heart Diseases; Cardiovascular Diseases; Atrial Fibrillation; Anti-Arrhythmia Agents
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Subjects undergoing cardiac surgery via complete median sternotomy
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Group 1: 20 subjects in the control group, which is the standard of care (i.e., no CardiaMend-Amioda (No Intervention): Subjects in treatment Group 1 (control) will receive no CardiaMend-Amiodarone patches.
- Group 2: 20 subjects receiving CardiaMend-Amiodarone infused with 70 mg of amiodarone (Experimental): Subjects in Group 2 (70 mg) will receive three patches each as follows:
  * One patch (5x6 cm) will be placed on top of the right atrium;
  * One patch (3x5 cm) will be placed within the transverse sinus near the dome of the left atrium; and
  * One patch (3x5 cm) will be placed within the oblique sinus on the posterior/inferior aspect of left atrium
  Interventions: Combination Product: The intervention includes Amiodarone-Infused CardiaMend patches (70mg, 150mg and 300mg)
- Group 3: 20 subjects receiving CardiaMend-Amiodarone infused with 150 mg of amiodarone. (Experimental): Subjects in Group 3 (150 mg) will receive three patches each as follows:
  * One patch (5x6 cm) will be placed on top of the right atrium;
  * One patch (3x5 cm) will be placed within the transverse sinus near the dome of the left atrium; and
  * One patch (3x5 cm) will be placed within the oblique sinus on the posterior/inferior aspect of left atrium
  Interventions: Combination Product: The intervention includes Amiodarone-Infused CardiaMend patches (70mg, 150mg and 300mg)
- Group 4: 20 subjects receiving CardiaMend-Amiodarone infused with 300 mg of amiodarone. (Experimental): Subjects in Group 4 (300 mg) will receive three patches each as follows:
  * One patch (5x6 cm) will be placed on top of the right atrium;
  * One patch (3x5 cm) will be placed within the transverse sinus near the dome of the left atrium; and
  * One patch (3x5 cm) will be placed within the oblique sinus on the posterior/inferior aspect of left atrium
  Interventions: Combination Product: The intervention includes Amiodarone-Infused CardiaMend patches (70mg, 150mg and 300mg)

INTERVENTIONS:
Combination Product: The intervention includes Amiodarone-Infused CardiaMend patches (70mg, 150mg and 300mg) — Intervention includes a topical, atrial-specific, amiodarone infused CardiaMend patch in the operating room and applied onto the epicardial surface biatrially
  Arms: Group 2: 20 subjects receiving CardiaMend-Amiodarone infused with 70 mg of amiodarone; Group 3: 20 subjects receiving CardiaMend-Amiodarone infused with 150 mg of amiodarone.; Group 4: 20 subjects receiving CardiaMend-Amiodarone infused with 300 mg of amiodarone.

SUMMARY:
The goal of this clinical trial is to is to test the safety of a new way to deliver a commonly used drug (amiodarone) used in heart surgery by placing a patch containing the drug directly on the heart instead of in an IV (vein). Participating subjects must be 20-85 year old males or females. Up to 80 participants having cardiac surgery at the University of Louisville will be involved in this study.

The main questions this study aims to answer are:

1. Is the patch safe?
2. Does the patch lower the rate of atrial fibrillation (irregular heart rhythm) after cardiac surgery?

Researchers will compare up to 3 different doses of the amiodarone patches (low, medium and high) to the usual treatment (Standard of Care) to see if there are differences (increases or decreases) in heart rhythms after cardiac surgery across study groups.

Participants will be placed in one of 4 study groups:

* Standard of Care (20 participants)
* Low dose patch (20 participants)
* Medium dose patch (20 participants)
* High dose patch (20 participants)

Participants will be monitored closely by their doctor(s) during the study and would:

* Agree to participate after having their doctor, or a member of the team, explain the study in detail and allowing them to ask any questions they would like.
* Sign an Informed Consent Form which will describe the study and tests in full.
* Agree to have their doctor and his/her research team record your medical information, draw blood, and perform electrocardiograms, or EKGs (quick, painless test that measures the electrical activity of the heart) and echocardiograms (image of heart) to monitor their heart.
* Agree to receive training on the portable EKG recorder and to use it at home approximately 30 days and 6 months after their surgery to monitor their heart.
* Agree to return to the hospital approximately 30 days and 6 months after their surgery for a study visit.

Participant involvement will be approximately 7 months total.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety of a drug-device treatment for the prevention of postoperative atrial fibrillation following open heart surgery. Approximately a quarter of patients will develop atrial fibrillation after open heart surgery. Atrial fibrillation is a type of irregular heart rhythm or arrhythmia, in which the heart does not pump effectively. This can lead to problems such as stroke, palpitations (an abnormal heart rhythm that can feel like your heart is racing or pounding) and prolonged hospital stays. The goal of this study is to determine if the application of a medication (amiodarone) containing patch on the surface of the heart at the time of surgery is safe, which may lead to a treatment to lower the rate of atrial fibrillation in patients undergoing open heart surgery. The study drug-device is not yet FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 20-85 years old.
* Subjects able to give voluntary written informed consent, who understand and are willing to comply with study-related procedures.
* Subjects scheduled to undergo open-chest cardiac surgery via complete median sternotomy.
* Subjects in sinus rhythm at the time of office visit and during prior EKG (note: continuous EKG monitoring for 48 hours is not required).

Exclusion Criteria:

* Subjects unable to give voluntary written informed consent, unlikely to cooperate, or legally incompetent, including subjects institutionalized by court or official order, or in a dependency relationship with testing center or investigator.
* Subjects with a condition that could interfere with their ability to comply with the study.
* Subjects participating in an interventional clinical study or who have participated in such study during the preceding 30 days.
* Female subjects who are pregnant, breastfeeding, were pregnant within the last three months, or are planning to become pregnant during the study.
* Subjects with active skin or deep infection at the site of implantation.
* Subjects with a history of chronic wounds or wound-healing disorders.
* Subjects with known connective tissue diseases (e.g. Ehlers-Danlos syndrome, Epidermolysis bullosa, Marfan syndrome, Osteogenesis imperfecta).
* Subjects who are Immune-suppressed or with immune deficiency (properly managed diabetes mellitus is not an exclusion criterion).
* Subjects on concomitant oral or IV systemic corticosteroid therapy and/or other constant anti-inflammatory therapies.
* Subjects on the following medications with known interactions with amiodarone: doxorubicin, fosphenytoin, lopinavir-ritonavir, ledipasvir/sofosbuvir, quinidine , procainamide, disopyramide, other Vaughan William class III agents including dofetilide, dronedarone, ibutilide and vernakalant.
* Subjects with coadministration of any medications which cause QT prolongation
* Subjects with implantable cardiac devices (i.e., cardiac resynchronization therapy devices with and without defibrillator capabilities (CRTs and CRT-Ds), implantable cardioverter-defibrillators (ICD), and pacemakers).
* Subjects with a known history of atrial fibrillation or paroxysmal atrial fibrillation.
* Subjects with a history of ablation for atrial fibrillation.
* Subjects already receiving amiodarone as a treatment for atrial fibrillation or ventricular arrhythmias.
* Subjects with a disease of the left pleura, previous intervention in the left pleural space, or chest deformity.
* Subjects with heart failure (BNP>1000), low ejection fraction (<35%), end-stage renal disease (on dialysis or GFR<20).
* Subjects electing to receive an ablative procedure for atrial fibrillation during the index operation.
* Subjects with prior cardiac surgery via sternotomy.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety, defined as major adverse cardiac and cerebrovascular events (MACCE), up to subject discharge. | From the day of the index procedure up to two months or date of hospital discharge, whichever is the sooner
  MACCE is defined as in-hospital all-cause death, acute myocardial infarction (AMI), or ischemic stroke.

SECONDARY OUTCOMES:
Incidence of postoperative atrial fibrillation (POAF) | From the day of the index procedure up to two months or date of hospital discharge, whichever is the sooner
  Incidence of POAF up to patient discharge; defined as subject experiencing atrial fibrillation/flutter (AF) after OR Exit that lasted longer than one hour, or lasted less than one hour but required medical or procedural intervention.
Migration of cardiamend-amiodarone patches. | One day before the date of hospital discharge up to two months
  Confirm placement of patches with non-contrast thoracic CT scan on first 3 subjects from Group 2 (70 mg) prior to discharge.
Length of Stay. | From the day of the index procedure to hospital discharge up to 2 months
  Length of initial hospital stay.
Hospital readmission. | Up to 30 days post-subject hospital discharge.
  30 day readmission from discharge due to all cause complications based upon STS data
POAF duration | From the day of the index procedure up to two months or date of hospital discharge, whichever is the sooner
  Duration of POAF, if observed.
Discharge on antiarrhythmic drug. | At subject hospital discharge to a maximum of 2 months post-index procedure date.
  Discharge on antiarrhythmic drug, if POAF observed.
Discharge on oral anticoagulation. | At subject hospital discharge to a maximum of 2 months post-index procedure date.
  Discharge on oral anticoagulation, if POAF observed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Slaughter, MD, Principal Investigator — University of Louisville Hospitals
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No